CLINICAL TRIAL: NCT01430273
Title: Assessment of Blood Loss With a Point Of Care Device During Hip/Knee Surgery Performed On Dual/Single Antiplatelet Therapy
Brief Title: Assessment of Blood Loss With a Point Of Care Device
Acronym: BLOOD
Status: Terminated | Type: Observational
Why Stopped: recruiting centers do not have the patient potential
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: NI10028; 2010-A01454-35 (Other: IDRCB)
Record Dates: First submitted 2011-08-04; First posted 2011-09-08 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Acute or Programmed Hip Replacement (Gamma Nail, Total Prosthesis or Throuhg DHS) / Knee Surgery
Keywords: Antiplatelet therapy; Surgery; Bleeding; Platelet aggregation
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — salivary kit (Oragnèe-DNA approved by FDA) or blood (2 tubes 2.5ml)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Planned hip or knee arthroplasty: Patients with planned hip or knee arthroplasty
- urgent hip or knee arthroplasty: Patients with hip or knee arthroplasty in emergency.

SUMMARY:
Main Objective: The purpose of this study is to demonstrate whether there is a correlation between perioperative blood loss and the degree of platelet inhibition assessed by a point of care assay in patients undergoing hip or knee arthroplasty and treated by antiplatelet mono/bi-therapy

DETAILED DESCRIPTION:
Type of study : Prospective, non-interventional, multicenter registry Principal Investigator: Collet Jean-Philippe Rational: Discontinuation of antiplatelet therapy in patients with established coronary artery disease (CAD) has become an increasingly important concern given the risk of recurrent arterial event. Exaggerated concern about increased procedure-related bleeding remains the major factor for premature discontinuation of APT. Interruption modalities and their impact on perioperative bleeding has never been prospectively evaluated and it is accepted that the maximum duration of interruption should not exceed 5 days for Clopidogrel/Ticagrelor and 7 days for Prasugrel given the fact that the remaining antiplatelet effect of APT is observed in less than 50% of patients after 3 days of interruption. Resuming APT after the operation has never been studied and remains a complex situation during anticoagulation is often prescribed to prevent deep vein thrombosis further increasing perioperative bleeding.

Hypotheses: (i) the volume of perioperative blood loss is correlated to the degree of platelet inhibition. (ii) Clopidogrel metabolizer status as defined by genetic profile is also correlated to perioperative blood loss. (iii) Resuming antiplatelet therapy during the perioperative period is not associated with a significant recovery of the antiplatelet effect.

Primary endpoint: Perioperative (day 1-day 5) blood loss in mL assessed by NADLER & Mercurial formula* and PRU** (for patients under Clopidogrel/ARU*** as measured using the VerifyNow®P2Y12 and aspirin assays at baseline. Secondary objectives: (i) to evaluate the correlation between clopidogrel genetic metabolizer status**** and perioperative blood loss. To evaluate antiplatelet pharmacodynamic response at discharge according to metabolizer status. Definition*Blood loss in mL of Red Blood Cell (RBC) = Compensated RBC Volume (1 Pack=150mL) + Non Compensated RBC Vol. (Total Blood Loss : Ht D-1-Ht D+5). *PRU=Platelet Reaction Unit. It is a specific measure of on-clopidogrel platelet reactivity. Cut-off value is for defining high-on clopidogrel platelet reactivity is 230. **ARU=Aspirin Reaction Unit. It is a specific measure of on-aspirin platelet reactivity. Cutoff value to identify high on-aspirin platelet reactivity is 550. ***Clopidogrel Metabolizer Phenotype is defined according to the carriage of the loss/gain-of function allele 2C19*2-*8/*17 as follows: SM for slow metabolizer: (*2-*8/*2-*8) ; Ultrafast Metabolizer (FM): (*17/*17) ; Normal/intermediate (M): (wt/wt, wt/*17, *2-*8/*17 or *2-*8/wt)

Number of subjects : 200 patients

Study duration: Two years.

Study duration per subject: length of hospital stay with a maximum duration of 30 days.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Patient in antiplatelet monotherapy (aspirin or clopidogrel) or dual therapy (aspirin + clopidogrel / prasugrel / ticagrelor) in the context of secondary prevention after:

  * acute coronary syndrome
  * and / or intracoronary stenting
* Planned or urgent hip (gamma nail, total prosthesis or through DHS) or knee arthroplasty
* Informed consent of the participant
* Patient receiving a social security scheme or entitled

Exclusion Criteria:

* Polytrauma
* Anemia <9g/dL
* Indication for oral anticoagulation
* Pelvic fracture justifying complex surgery
* Ongoing or recent major bleeding or recent major surgery (< 3 weeks)
* Liver failure
* Thrombopenia <80 000/µl
* Lack of health insurance
* Mental disability
* Participation to any other research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets CAD patients exposed to antiplatelelt mono/bitherapy who need planned or emergency knee/hip athroplasty. This innovative study will bring new insights on how works antiplatelet therapy during the perioperative period according to drug exposition and metabolizer profile.
  Patients ethnicity will be recorded and defined according to the place of birth of the participants and of their parents given the identification of the metabolizer profile with respect to the CYP 2C19*2 carriage. The analysis will bestratified according to ethnicity to avoid biases.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss in mL assessed by NADLER & Mercurial formula* and PRU**/ARU*** as measured using the VerifyNow®P2Y12 and aspirin assays at baseline | day 1- day 5
  Perioperative (day 1-day 5) blood loss in mL assessed by NADLER & Mercuriali formula* and PRU**/ARU*** as measured using the VerifyNow®P2Y12 and aspirin assays at baseline.

SECONDARY OUTCOMES:
Evaluate the correlation between clopidogrel genetic metabolizer status**** and perioperative blood loss. | up to 10 days
  When the patient discharges of surgery department
To evaluate clopidogrel and aspirin pharmacodynamic response at discharge according to metabolizer status. | up to 10 days
  When the patient discharges of surgery department

CONTACTS AND LOCATIONS:
Overall Officials: COLLET Jean-Philippe, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Institute of cardiology - Pitié Salpêtrière Hospital, Paris
  - pôle Anesthesie -Réanimation- CHU Pitie -Salpetrière, Paris
  - CHU Toulouse - Hôpital de Rangueil - Anésthésie-Réanimation, Toulouse